CLINICAL TRIAL: NCT03801187
Title: Surgical Protocol for Peri-implantitis in Horizontal Defect With Keratinised Tissue Using Er:YAG Laser or an Air-abrasive Device in Addition to Chlorhexidine: a Randomized Clinical Trial
Brief Title: Surgical Protocol for Peri-implantitis Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Marco Clementini, Principal Investigator, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: peri-implant surgical-1
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Peri-implantitis
Keywords: peri-implantitis; surgical treatment; Er:Yag laser; Air-flow; chlorhexidine
MeSH Terms: conditions — Peri-Implantitis | interventions — Chlorhexidine; Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chlorhexidine (Sham Comparator): Access flap will be raised to gain access to the implant surface. Inflammatory tissue, excess cement or plaque deposits will be removed using titanium curettes and the implant surface will be cleaned by copious irrigation with sterile saline and surgical gauze soaked in Chlorhexidine.
  Interventions: Procedure: chlorhexidine
- Er:YAG laser (Experimental): Er: Yag laser treatment will be provided on the implant surface.
  Interventions: Procedure: chlorhexidine; Procedure: Er:YAG laser
- Air Powder (Active Comparator): An Air-Powder treatment will be provided on the implant surface
  Interventions: Procedure: chlorhexidine; Procedure: Air-Powder

INTERVENTIONS:
Procedure: chlorhexidine — Inflammatory tissue, excess cement or plaque deposits will be removed using titanium curettes and the implant surface will be cleaned by copious irrigation with sterile saline and surgical gauze soaked in chlorhexidine.
Procedure: Er:YAG laser — Er.YAg laser treatment will be provided on the implant surface.
  Arms: Er:YAG laser
Procedure: Air-Powder — An air powder device will be treatment will be provided on the implant surface.
  Arms: Air Powder

SUMMARY:
Peri-implant diseases are common post-restorative complications in implant rehabilitations and they occur with an incidence of 12-43%.

Based on the available data in literature, the surgical therapy for peri-implantitis is effective in disease resolution. Surgical access to peri-implant lesions facilitates the removal of all granulation tissue from the defect area as well as debridement and decontamination of the exposed implant surface defect area.

Different techniques have been used for implant surface decontamination during peri-implant surgery, including mechanical, chemical and laser treatments.

DETAILED DESCRIPTION:
Peri-implantitis are defined as inflammatory diseases caused by bacterial biofilm around implant surface characterized by bleeding on probing, probing depth and eventually bone loss; if not successfully treated they may lead to implant loss. Based on the available parameters that have been reported in literature non surgical therapy doesn't seem to be effective on peri-implantitis. Therefore it is recommended to consider advanced therapies such as surgical interventions when non surgical peri-implant therapy fails to achieve significant improvements in clinical parameters.

Numerous approaches have been used for implant surface decontamination during peri-implant surgery, including mechanical, chemical and laser treatments.

Conventional mechanical means don't seem to be effective on peri-implant diseases. In addition, the rough implant surface is a retentive factor for bacterial colonization and therefore makes implant surface difficult to debride.

A treatment protocol that may offer an advantage over traditional mechanical treatment includes the use of laser therapy and air-powder devices. Data have shown that treatments with Er.Yag laser have a bactericidal effect and are safe and effective on implant surfaces. Slightly better clinical results in terms of debridement, probing depth, bleeding on probing and clinical attachment level have been reported by Er:Yag laser treatment compared with traditional non surgical mechanical debridement with titanium curettes and pellet with saline in the surgical treatment of peri-implantitis.

The air abrasive method for debridement has also been used on implant surfaces demonstrating no relevant adverse effect. Until now, powders based on sodium bicarbonate and glycine have been used with pressured air/water. Nowadays a less abrasive method involves the use of erythritol powder.

The aim of the present randomized controlled clinical trial is to assess the efficacy in improving clinical parameters of two further methods of implant decontamination (er:Yag laser or air-abrasive device) after chemical treatment and chemical cleaning during surgical treatment of peri-implantitis in addition to chlorhexidine in horizontal defects with keratinised tissue around implant surfaces.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least one screw-type titanium implant exhibiting bleeding and/or suppuration on probing combined with:

  1. PPD ≥ 5 mm and bone loss ≥ 2 mm (compared to crestal bone levels at the time of placement of the reconstruction)
  2. PPD ≥6 and bone loss ≥3 (not compared to crestal bone levels at the time of placement of the reconstruction)
* single tooth and bridgework restorations without overhangs
* no evidence of occlusal overload (i.e. occlusal contacts revealed appropriate adjustment),
* treated chronic periodontitis and proper periodontal maintenance care
* FMPS < 20%
* non-smoker or light smoking status in smokers (<10 cigarettes per day)
* implant function time ≥ 1 year.

Exclusion Criteria:

* Patients with uncontrolled diabetes
* patients with osteoporosis or under bisphosphonate medication,
* pregnant or lactating women
* patients with a history of radiotherapy to the head and neck region
* hollow implants
* implant mobility
* implants at which no position could be identified where proper probing measurements could be performed;
* previous surgical treatment of the peri-implantitis lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing changes | baseline, 3, 6 and 12 months after treatment
  changes of bleeding on probing, evaluated as present if bleeding will be evident within 30 s after probing, or absent, if no bleeding will be noticed within 30 s after probing,

SECONDARY OUTCOMES:
clinical attachment level changes | baseline, 3, 6 and 12 months after treatment
  changes in clinical attachment level, measured from CEJ to the tip of the probe
probing pocket depth changes | baseline, 3, 6 and 12 months after treatment
  changes in probing depth probing, measured from gingival margin to te tip of the probe
mucosal recession changes | baseline, 3, 6 and 12 months after treatment
  changes in mucosal recession, measured from CEJ to gingival margin
bone level changes | baseline and 12 months after treatment
  changes in bone level at mesial and distal aspect, measured on periapical X-ray

CONTACTS AND LOCATIONS:
Overall Officials: Massimo De Sanctis, Prof., Study Chair — Università Vita-Salute San Raffaele
Locations (1):
- Università Vita-Salute San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided